CLINICAL TRIAL: NCT03072394
Title: Anesthetic Ointment vs Local Injectable Anesthetic in Trans-radial Cardiac Catheterization: The RAOLA Study
Brief Title: Local Anesthesia in Radial Catheterization
Acronym: RAOLA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hippocration General Hospital (Other)
Responsible Party: Principal Investigator, Dimitris Tousoulis, Professor of Cardiology, Hippocration General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HippocratioGH
Record Dates: First submitted 2017-02-24; First posted 2017-03-07 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Anesthesia, Local; Coronary Artery Disease; Catheter Site Discomfort; Catheter Site Pain
MeSH Terms: conditions — Coronary Artery Disease | interventions — Anesthetics, Local; Anesthesia, Local

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMLA anesthetic ointment (AO) (Experimental): In AO group a layer of 2.5 gr EMLA cream (standard adult dose) is applied to both wrists, 1 cm above the styloid process of the radius 30 minutes before the puncture, by an experienced cathlab nurse.
  Interventions: Drug: Local anesthetic
- Local Skin Anesthetic Injection (LA) (Active Comparator): In LA group the radial artery is infiltrated with 1-2 mL of 2% lidocaine, using a 26 G needle, 0.5-1 cm proximal to the styloid process one minute before the puncture
  Interventions: Drug: local anaesthetic injection

INTERVENTIONS:
Drug: Local anesthetic — Local skin anesthesia during radial coronary artery catheterization by EMLA anesthetic ointment
  Other Names: Local anesthetic ointment
  Arms: EMLA anesthetic ointment (AO)
Drug: local anaesthetic injection — Local skin anesthesia during radial coronary artery catheterization by lidocaine injection
  Other Names: Skin anethesia by lidocaine injection
  Arms: Local Skin Anesthetic Injection (LA)

SUMMARY:
A randomized clinical trial to test the efficacy of EMLA cream (lidocaine 2.5% and prilocaine 2.5% in a ratio of 1:1 by weight) in comparison to the established local anesthesia (LA) protocol of lidocaine subcutaneous injection, in providing adequate peri-operative local anesthesia during transradial coronary angiography.

DETAILED DESCRIPTION:
A total of 444 consecutive patients, who are referred for elective coronary angiography to 1st Cardiology Department cathlab, with the suspicion of coronary artery disease (CAD) will be enrolled in this study. Exclusion criteria are acute coronary syndrome, previous ipsilateral transradial approach, Raynaud's syndrome, abnormal renal function with or without need for hemodialysis, known history of sensitivity to local anesthetics, non-palpable radial pulse, abnormal Barbeau's test and patient's refusal. Baseline clinical, demographic and procedural data of the study population were recorded.

Participants will be randomly assigned to either the EMLA (AO) or the lidocaine group (LA), by a randomization table.

Primary end-point: the perception of radial pain assessed during artery puncture and 30 minutes after sheath removal.

Secondary end-point: The number of puncture attempts, the total time required before successful sheath insertion, and the occurrence of radial artery spasm will be also documented in each group

Participants will be observed for 4 hours post angiography for development of local complications or side effects.

ELIGIBILITY:
Inclusion Criteria:

* referral for elective diagnostic coronary angiography

Exclusion Criteria:

* acute coronary syndrome, previous ipsilateral transradial approach, Raynaud's syndrome, abnormal renal function with or without need for hemodialysis, known history of sensitivity to local anesthetics, non-palpable radial pulse, abnormal Barbeau's test and patient's refusal.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2015-01-10 (Actual); Primary Completion 2020-11-20 (Estimated); Study Completion 2021-01-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale of Pain Perception during sheath insertion | During artery puncture
  The primary end-point of the study is the perception of radial pain assessed during artery puncture
Visual Analog Scale of Pain Perception after sheath removal | 30 minutes after sheath removal
  The primary end-point of the study is the perception of radial pain assessed 30 minutes after sheath removal

SECONDARY OUTCOMES:
Puncture efficiency (number of puncture attempts) | During radial artery catheterization
  The number of puncture attempts, the total time required before successful sheath insertion are documented in each group and constitute the secondary end points of the study.
Radial artery spasm | During radial artery catheterization
  The occurrence of radial artery spasm in each group during radial artery catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Tousoulis, MD PhD, Study Director — Professor of Cardiology; George Latsios, MD PhD, Principal Investigator — Consultant Cardiologist
Locations (1):
- Hippocration Hospital, Athens University Medical School, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No